CLINICAL TRIAL: NCT03168243
Title: Evaluating the Tolerance, Compliance and Acceptability of a Nutritionally Complete, High Energy, High Protein, Enteral Feed in Adults - a Pilot Study
Brief Title: High Energy High Protein Tube Feed Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NPPE001
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Nutrition
Keywords: nutrition support, home enteral feeding

STUDY DESIGN:
Intervention Model Description: This is a prospective, single arm, longitudinal, interventional, multi-centre study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Energy High Protein Tube Feed (Experimental): As study is a single arm design, all patients will be in the intervention group. The will act as their own control by means of a 3 day baseline period. All patients in the study will receive the same intervention, the high energy high protein tube feed, in quantities specified by their dietitian based on their nutritional requirements.
  Interventions: Dietary Supplement: High Energy High Protein Tube Feed

INTERVENTIONS:
Dietary Supplement: High Energy High Protein Tube Feed — Following a 3 day baseline period all patients will receive the high energy, high protein tube feed for a period of 4 weeks (28 days).

SUMMARY:
Enteral tube feeds are commonly used to meet the entire or partial nutritional requirements of patients with disease-related malnutrition and other conditions who need nutrition support. A large proportion of tube fed patients have increased protein and/or energy requirements due to a higher body mass or increased metabolic stress as a result of disease, surgery or trauma. A high energy, high protein feed has been developed to help meet the needs of such patients. The aim of this study is to investigate the tolerance, compliance and acceptability of this high energy high protein tube feed in adult patients who require nutritional support via tube feeding. 50 eligible patients requiring tube feeding will receive the high energy, high protein feed, according to nutritional requirements for 4 weeks. The primary outcome is nutritional intake, and secondary outcomes include gastrointestinal (GI) tolerance, compliance, acceptability and functional measures. Additional exploratory outcomes of quality of life and micronutrient levels will also be investigated.

DETAILED DESCRIPTION:
Introduction

The present study will investigate the effect of a high energy, high protein tube feed in patients requiring enteral feeding in the community. The primary objective is to evaluate the effect of daily intake of the high energy, high protein tube feed, in addition to appropriate nutritional management, on total nutrient intakes for 4 weeks. The secondary objectives are to evaluate the effect of daily intake of the feed on gastrointestinal tolerance, compliance, acceptability and functional measures. Additional exploratory measures will be quality of life and micronutrient levels. Enteral tube feeding patients will be recruited by the dietitians responsible for their care, from a variety of dietetic services across the United Kingdom. Potential participants that require a high energy, high protein tube feed will already be known to the Investigating Dietitian or dietetic team at the investigating sites or will be referred to the dietetic service during the duration of the study.

Intervention

Following a 3 day baseline period, each patient will receive the high energy, high protein tube feed for a period of 4 weeks (28 days). The appropriate feed and prescription will be determined on an individual basis by the Dietitian responsible for the patient's nutritional management, based on the patient's clinical requirement and preference and the Dietitian's clinical judgement.

The study feed is classed as a 'Dietary Food for Special Medical Purposes' (EC Directive 1999/21/EC, 1999).

Outcome measures

1. Nutrient intake (energy, protein, fluid and micronutrients)
2. Gastro-intestinal tolerance Gastro-intestinal tolerance will be measured using a standardised gastro-intestinal tolerance questionnaire.
3. Compliance with feed prescription Compliance with feed prescription will be assessed daily throughout the study
4. Acceptability Feed acceptability, such as preference and ease of use will be assessed at the end of study.
5. Anthropometry Weight and height will be measured where possible using standard measures.
6. Patient history Previous nutritional support provided to the patient, previous enteral feeding products prescribed, history of intolerance, the need for a high energy, high protein feed, weight history and other relevant dietetic history.
7. Muscle Function (Hand Grip Strength)
8. Quality of life
9. Micronutrients levels

Statistical aspects

As this is a pilot study no power calculation was undertaken. The sample size of this trial is similar to other published trials of tube feeds in patient populations. In addition to helping to inform clinical practice, the data collected will also be used to support an application to the Advisory Committee of Borderline Substances (ACBS). Recruiting a sample of 50 patients should enable sufficient data to be collected to meet ACBS requirements for the study, while allowing for drop outs during the study period.

Data will be analysed using repeated measures analysis of variance (ANOVA) or t-test where appropriate. Categorical data will be analysed using appropriate methods (e.g. chi-squared). Interim analysis may be undertaken after 30 patients have been recruited. Statistical analysis will be undertaken using IBM SPSS version 23.0 Armonk, New York, USA.

Ethical Considerations

This study will be undertaken in adults with capacity to consent only. In line with the guidance of the Medical Research Council, written informed consent will be obtained for each participant taking part in the study. The investigator will ensure that the study will be conducted in full conformance with the principles of the 'Declaration of Helsinki' (64th WMA General Assembly, Fortaleza, Brazil, October 2013) and with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the individual.

Study Monitoring

Monitoring will be organised by the sponsor to evaluate the progress of the study, verify the accuracy and completeness of the Case Report Forms (CRFs) and to ensure adherence to the protocol. Monitoring visits will be scheduled periodically in consultation with the investigator. During monitoring, the study monitor will need access to all patient's study records and raw data used for and generated during the study needed to verify the data in the CRF. If necessary, the investigator must provide the monitor any required background data.

Confidentiality

On recruitment to the study, all participants will be allocated a unique study number, which will be the only identifier on all participant data that will leave the institution involved. For patients consenting to provide blood samples, names will be required to be stored with blood sample results. These results will be accessible by the Investigating Dietitian responsible for the patient's care. For the purposes of data analysis and any publication and dissemination of the data, all results will be analysed and identified using the patient's unique study number only. No identifiable personal data will be published.

ELIGIBILITY:
Inclusion Criteria

* Male or female
* Age 18 years and over
* Requiring tube feeding in the community to meet nutritional requirements
* Expected to receive at least 500kcal from tube feeding
* Capacity to consent

Exclusion Criteria

* Patients receiving parenteral nutrition
* Patients with major hepatic dysfunction (i.e. decompensated liver disease)
* Patients with major renal dysfunction (i.e. requiring filtration or Stage 4/5 chronic kidney disease (CKD))
* Patients in intensive care
* Patients with galactosaemia or severe lactose intolerance
* Participation in other clinical studies within 2 weeks prior to entry of this study
* Inability to provide informed consent
* Investigator concern around willingness/ability of patient to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change in nutrient intakes (energy, protein, fluid and micronutrients) | Measurements will be taken at Baseline (DAY 1) and End of Study (DAY 31).
  Nutrient intakes, including the intake of all nutrition provided (including the study feed, other enteral tube feeding, foods, drinks and oral nutritional supplements) will be recorded using 24hr diet recalls. Nutritics® (https://www.nutritics.com/p/references), a dietary analysis program, will be used to calculate energy, protein, micronutrient and fluid intakes.

SECONDARY OUTCOMES:
Gastro-intestinal tolerance | Gastro-intestinal tolerance will be recorded at baseline (DAY 1, 2 and 3) and on days 4, 5, and 6 of the study (the first 3 days the patient is taking the study feed) and once at the end of each week the patient is taking the feed.
  Tolerance will be recorded using a standardised gastro-intestinal tolerance questionnaire, measuring incidence and severity of gastro-intestinal symptoms and Bristol Stool Chart© type and frequency of bowel movements, to be completed by the patient.
Compliance with feed prescription measured via daily feed intake recoding | Every day throughout study completion, 31 days in total.
  Compliance will be assessed daily throughout the Baseline period and Intervention period by recording how much study feed was received, to be recorded by the patient or carer. The amount prescribed by the Dietitian will be recorded at the start of the study, and any changes to this prescription also noted. Compliance will be calculated as feed taken as a percentage of feed prescribed.
Acceptability | End of study (DAY 31)
  Feed acceptability (preference, ease of use) will be assessed at the end of study by a questionnaire completed by the patient or carer.
Muscle Function (hand grip strength) | Measurements will be taken at Baseline (DAY 1) and End of Study (DAY 31).
  Hand grip strength will be measured, where possible, in all patients in the dominant arm using a handgrip dynamometer. Three measurements will be taken and the mean used for analysis.
EQ-5D Quality of life | Measurements will be taken at Baseline (DAY 1) and End of Study (DAY 31).
  Quality of life will be measured using the EQ-5D questionnaire.
Micronutrient status | Measurements will be taken at Baseline (DAY 1) and End of Study (DAY 31).
  In a subset of patients blood samples will be taken and analysed to assess micronutrient status.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, PhD, Principal Investigator — Nutricia Ltd
Locations (7):
- United Kingdom (7):
  - Lewisham Health Care NHS Trust, Lewisham, London
  - Somerset Partnership NHS Foundation Trust, Bridgwater, Somerset
  - Western Sussex Hospitals NHS Trust, Worthing, West Sussex
  - University Hospitals Bristol, Bristol
  - Aneurin Bevan University Health Board, Caerleon
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No